CLINICAL TRIAL: NCT00568243
Title: Visual Motor Coordination
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080031; 08-EI-0031
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteer; Neurodegenerative Diseases
Keywords: Visuomotor Integration; Visual Attention; Eye Movements; Reaction Time; Natural History; Saccades; Healthy Volunteer; HV
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Volunteer: Healthy subjects without neurodegenerative diseases
- Patients: Subjects with neurodegenerative diseases

SUMMARY:
Background:

* The relation between eye movement and brain function is a subject of interest to the National Eye Institute.
* By comparing eye movement in healthy volunteers to research conducted on patients who have difficulty moving their eyes, the National Eye Institute hopes to develop and improve diagnostic procedures for people with eye diseases.

Objectives:

-The purpose of this study is to understand how we see visual patterns and how we move our eyes to see.

Eligibility:

* Normal volunteers:

  * must have no serious illnesses and must be 18 years of age or older
  * are able to follow directions and pay attention to visual stimuli and respond as appropriate
  * individuals with a history of eye or brain diseases, or previous eye or eye muscle surgery, are not allowed to participate in this study. Individuals who are currently using eye medications also are not eligible for the study.
* Patients:

  * who are 18 years of age or older
  * are able to follow directions and pay attention to visual stimuli and respond as appropriate

Design:

* Participants will visit the National Eye Institute outpatient clinic for examination and testing.
* Participants will be screened with a medical history and eye examination (including eye pressure and eye movement tests).
* Participants with healthy eyes will participate in eye movement testing experiments:

  * One or more sessions lasting less than three hours each.
  * Eye movements will be recorded with a video/infrared camera system.
  * For the majority of the studies done under this protocol, only one or two sessions will be required. A few studies recording very small eye movements will require three or more sessions.

DETAILED DESCRIPTION:
Study Description: This natural history study will investigate eye movements and other responses to visual stimuli in normal individuals (normal volunteers) and patients. Normal adult volunteers will be recruited and will undergo an eye exam to assure that there are no visual system problems. . Volunteers will be studied in one or more sessions where eye movement, verbal, or hand movement responses are recorded in response to visual stimuli. Patients with diseases affecting the oculomotor or visual systems will also be recruited to help us better understand these systems and to help characterize their specific disease.

Objectives:

The objective is to study normal volunteers and patients for eye movement and other responses to visual stimuli with the goal of better understanding human vision and neural control of eye movements.

Endpoints:

The primary outcome measure is eye movement and other responses to visual stimuli.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Normal Volunteers:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Participant must be a volunteer with no ocular, visual, or oculomotor problems.
2. Participant must be 18 years old or older.
3. Participant must be able to follow directions and actively pay attention to visual stimuli and respond as appropriate.
4. For studies which use the contact lens, participant must be able to tolerate a contact lens in either one or both eyes.

Inclusion Criteria for Patients:

In order to be eligible to participate in this study, an individual must meet all of the following criteria

1. Participant must be 18 years old or older.
2. Participant must be able to follow directions and actively pay attention to visual stimuli and respond as appropriate.
3. For studies which use the contact lens, participant must be able to tolerate a contact lens in either one or both eyes.

EXCLUSION CRITERIA:

Exclusion Criteria for Normal Volunteers:

An individual who meets any of the following criteria will be excluded from participation in this

study:

An individual who meets any of the following criteria will be excluded from participation in thisstudy:

1. Participant has a history of ocular or visual diseases or diseases affecting the nervous system (including myasthenia, MS, etc.) or any diseases which might affect control of eye movements or affect vision.
2. Participant has had prior eye or eye muscle surgery.
3. Participant has a history of eye patching (amblyopia or lazy eye).
4. Participant currently uses eye drops or ocular medications.

Exclusion Criteria for Patients:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patient is unable to cooperate with testing, including sitting still while eye movements are recorded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal adult volunteers and patients with eye movement problems including strabismus or neuro-degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-12-04 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
eye movement/responses to visual stimuli | one to many times depending if normal volunteer or patient and the number of trials required to achieve clean data for small eye movements.
  Analysis of eye movements to characterize basic processes (normal volunteers) and to judge disease progress (in patients)

CONTACTS AND LOCATIONS:
Overall Officials: Rich J Krauzlis, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
.The raw data is eye movement tracings which are of no utility except in the context of a study with multiple subjects. Obtained results will be published and if requested, original data will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-EI-0031.html